CLINICAL TRIAL: NCT04257084
Title: A Multicenter, Randomized Controlled Trial for Surveillance in Ulcerative Colitis: Narrow Band Image Versus Chromoendoscopy for High-risk Groups
Brief Title: Surveillance in Ulcerative Colitis: Narrow Band Image Versus Chromoendoscopy for High-risk Groups
Acronym: SUNRISE-High
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Yonsei University (Other); Samsung Medical Center (Other); Sungkyunkwan University (Other); Ewha Womans University (Other); The Catholic University of Korea (Other); Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Dong-Hoon Yang, Clinical Associate Professor, Asan Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: SUNRISE-High
Record Dates: First submitted 2020-02-02; First posted 2020-02-05 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Ulcerative Colitis; Dysplasia
Keywords: chromoendoscopy; narrow band image; surveillance
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Narrow Band Imaging

STUDY DESIGN:
Intervention Model Description: a randomized controlled crossover trial
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CE-NBI (Active Comparator): High definition chromoendoscopy with target biopsy, at 1st surveillance colonoscopy during the trial High definition NBI with target biopsy, at 2nd surveillance colonoscopy during the trial
  Interventions: Diagnostic Test: chromoendoscopy with target biopsy; NBI with target biopsy
- NBI-CE (Active Comparator): High definition NBI with target biopsy, at 1st surveillance colonoscopy during the trial High definition chromoendoscopy with target biopsy, at 2nd surveillance colonoscopy during the trial
  Interventions: Diagnostic Test: chromoendoscopy with target biopsy; NBI with target biopsy

INTERVENTIONS:
Diagnostic Test: chromoendoscopy with target biopsy; NBI with target biopsy — Chromoendoscopy with target biopsy: 0.03% indigo carmine solution based chromoendoscopy (using high-definition colonoscopy) will be fulfilled and target biopsies will be taken at all abnormal mucosal lesions suspected dysplasia/neoplasia.
  NBI with target biopsy: After inserting a high definition colonoscopy up to cecum, endoscopists observe the colon in combination of white light and NBI (white light first and then NBI). Target biopsies will be taken at all abnormal mucosal lesions suspected dysplasia/neoplasia.

SUMMARY:
The risk of colorectal cancer (CRC) is increased in patients having ulcerative colitis (UC). Patients with long-standing extensive colitis, concomitant primary sclerosing cholangitis, or previous history of dysplasia carry an exceptionally high risk of CRC and require regular and short-interval surveillance colonoscopy. Recent guidelines recommend surveillance colonoscopy based on target biopsy rather than random biopsy applying chromoendoscopy (CE) or narrow band image (NBI) technique in UC at risk for CRC. However, the diagnostic yield of NBI-based surveillance and CE-based surveillance is not extensively investigated in the high-risk UC population. The investigators aimed to compare the dysplasia detection rate of NBI with that of CE in UC patients with a high risk of CRC by performing a multicenter, randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* At least one of the followings should be satisfied;

  1. A patient having extensive ulcerative colitis with 8-year or longer disease duration
  2. A patient having both ulcerative colitis and primary sclerosing colitis
  3. A patient having a previous history of dysplasia at the colitic segment within recent 5 years

Exclusion Criteria:

* All of the following conditions should be excluded for 1st surveillance colonoscopy study

  1. A patient who underwent total or segment colectomy.
  2. A patient who taking (warfarin or direct oral anticoagulants and cannot stop them for procedures owing to the high thromboembolic risk
  3. A patient who has known thrombocytopenia (less than 80,000/µL in recent 6 months
  4. A patient who has a coagulopathy
  5. A patient who has chronic renal disease evidenced by serum creatinine > 1.2 mg/dL within 6 months of study participation
  6. A patient who has already undergone surveillance colonoscopy within 1 year
* All of the following conditions should be excluded for 2nd surveillance colonoscopy study even if they were included in 1st surveillance study.

  1. A patient who underwent total or segment colectomy after 1st surveillance colonoscopy for this trial.
  2. A patient who taking (warfarin or direct oral anticoagulants and cannot stop them for procedures owing to the high thromboembolic risk
  3. A patient who has known thrombocytopenia (less than 80,000/µL in recent 6 months
  4. A patient who has a coagulopathy
  5. A patient who has chronic renal disease evidenced by serum creatinine > 1.2 mg/dL within 6 months of study participation

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Dysplasia detection rate at first surveillance | 3 months after first surveillance colonoscopy in each arm
  Any dysplasia within the colitic segments will be counted as "dysplasia" to calculate dysplasia detection rate. A sessile serrated lesion (SSL) with dysplasia located in the colitic segment will be counted as "dysplasia", but SSLs without dysplasia will not be counted as "dysplasia" even if located within colitic segments.
Neoplasia detection rate at first surveillance | 3 months after first surveillance colonoscopy in each arm
  Neoplasia at any segments (regardless of colitis) will be counted as "neoplasia" to calculate neoplasia detection rate. SSL will be counted as neoplasia
Dysplasia detection rate at second surveillance | 3 months after second surveillance colonoscopy in each arm
  Any dysplasia within the colitic segments will be counted as "dysplasia" to calculate dysplasia detection rate. A sessile serrated lesion (SSL) with dysplasia located in the colitic segment will be counted as "dysplasia", but SSLs without dysplasia will not be counted as "dysplasia" even if located within colitic segments.
Neoplasia detection rate at second surveillance | 3 months after second surveillance colonoscopy in each arm
  Neoplasia at any segments (regardless of colitis) will be counted as "neoplasia" to calculate neoplasia detection rate. SSL will be counted as neoplasia

SECONDARY OUTCOMES:
SSL detection rate | 3 months after overall surveillance colonoscopy in each arm
  Whether located at colitic or non-colitic segments, SSL will be included for calculating SSL detection rate in each arm. Serrated epithelial changes (serrated epithelial changes in histology, but nor discrete border under colonoscopy or no dysplasia under microscopy) will not be considered as SSL.
Total procedure time | 3 months after overall surveillance colonoscopy in each arm
  The whole colonoscopy procedure time
Withdrawal time | 3 months after overall surveillance colonoscopy in each arm
  Time spent for withdrawal after excluding time for taking biopsies
Endoscopic features of target-biopsied lesions | 3 months after overall surveillance colonoscopy in each arm
  Pit and vascular patterns, Modified Paris classification (suggested by SCENIC group)
Procedure-related adverse events | 3 months after overall surveillance colonoscopy in each arm
  bleeding requiring hemostasis or transfusion, perforation, exacerbation of UC requiring admission (within 3 months after surveillance colonoscopy)

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Hoon Yang, MD, PhD, Principal Investigator — Asan Medical Center